CLINICAL TRIAL: NCT05154864
Title: The Optimal Ultrafiltration Protocol in Pediatric Cardiac Surgery: An Observational Cohort Study
Brief Title: Ultrafiltration in Pediatric Cardiac Surgery: An Observational Cohort Study
Status: Completed | Type: Observational
Sponsor: IWK Health Centre (Other)
Responsible Party: Principal Investigator, Dr. David Horne, Congenital Cardiac Surgeon, IWK Health Centre
Other Study IDs: 1024869
Record Dates: First submitted 2021-11-08; First posted 2021-12-13 (Actual); Last update posted 2022-01-03 (Actual); Status verified 2021-12

CONDITIONS: Congenital Heart Disease; Inflammation
MeSH Terms: conditions — Heart Defects, Congenital; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Patient plasma samples and ultrafiltrate effluent samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SBUF-SMUF: All patients underwent standard of care cardiac surgery, cardiopulmonary bypass and SBUF-SMUF with effluent removal of 30 ml/kg/hr and physiologic solution replacement of 25ml/kg/hr.
  Interventions: Procedure: SBUF-SMUF

INTERVENTIONS:
Procedure: SBUF-SMUF — Intra-operative continuous ultrafiltration

SUMMARY:
Infants and children undergoing cardiac surgery with cardiopulmonary bypass (CPB) can experience systemic inflammation that prolongs post-operative recovery. Ultrafiltration is an intra-opreative technique that is hypothesized to extract circulating inflammatory mediators during the CPB time. There have been only a few small studies looking at a limited number of inflammatory marker profiles in this context. Our institution uses an innovative form of ultrafiltration "subzero-balance simple-modified ultrafiltration" (SBUF-SMUF) throughout the entire CPB time. SBUF-SMUF has been our standard of care for the last 5 years. This observational seeks to describe the clinical and immunologic outcomes of infants and children undergoing cardiac surgery with CBP and SBUF-SMUF.

ELIGIBILITY:
Inclusion Criteria:

* Congenital cardiac patients (< 30kg) that have been consented to a planned cardiac surgery procedure requiring cardiopulmonary bypass at the IWK Health Centre.
* Patient or family consent to participate in the study.

Exclusion Criteria:

* Patient or family refusal to participate.
* Known genetic syndrome with multi-organ abnormalities and immune dysfunction such as DiGeorge Syndrome, Trisomy 18 or 13, Noonan syndrome.
* Known immunodeficiency syndrome or bone marrow pathology.
* Severe liver disease with abnormal synthetic liver function tests.

Max Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants and children less than 30kg undergoing cardiac surgery with cardiopulmonary bypass and subzero-balance simple modified ultrafiltration (SBUF-SMUF).
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Inflammatory Mediator Analysis | Plasma and ultrafiltrate effluent at pre-specified time points: Pre-Sternotomy (20min), Post-Sternotomy (30 min), every 30 minutes during cardiopulmonary bypass, 0 hours post-ultrafiltration, 12 hours post-ultrafiltration, 24 hours post-ultrafiltration
  Change in Concentrations of C1q, C2, C3, C3b, C4, C4b, C5, complement factor B, complement factor H, complement factor IC5a, CCL2 ,CCL3, CCL4, CCL5 (RANTES), CXCL1, CXCL2, CXCL10, GM-CSF, IL-1α, IL-1β, IL-1Ra, IL-2, IL-6, CXCL8 (IL-8), IL-10, IL-12 (p70), IL-17/IL-17A, IL-33, TNF (TNF-α), TRAIL, IFN-γ, E-Selectin, L-Selectin, P-Selectin, ICAM-1, VCAM-1, ET1.

SECONDARY OUTCOMES:
Vasoactive-Ventilation-Renal (VVR) Score | Pre-specified time points: ICU admission, 12,24,48,72,96,120 hours post-ultrafiltration.
  Scale 0-60
Vasoactive-Inotrope Score (VIS) | Pre-specified time points: ICU admission, 12,24,48,72,96,120 hours post-ultrafiltration.
  Scale 0-40
Ventilation Index (VI) | Pre-specified time points: ICU admission, 12,24,48,72,96,120 hours post-ultrafiltration.
  Scale 0-40
Oxygenation Index (OI) | Pre-specified time points: ICU admission, 12,24,48,72,96,120 hours post-ultrafiltration.
  Scale 0-20
Ventilation Time | Through study completion, an average of 1 week.
Intensive Care Unit Length of Stay | Through study completion, an average of 1 week.
  Standardized Discharge Criteria
Acute Kidney Injury | Through study completion, an average of 1 week.
  Kidney Disease Improving Global Outcomes criteria with Stages 1-3

OTHER OUTCOMES:
Arterial Blood Gas | Pre-specified time points: Pre-Sternotomy (20min), Post-Sternotomy (30 min), every 30 minutes during cardiopulmonary bypass, 0,12,24,48,72,96,120 hours post-ultrafiltration.
Red Blood Cell Transfusion | Measured through 24-hours post-operative
  volume in ml/kg
Plasma Transfusion | Measured through 24-hours post-operative
  volume in ml/kg
Platelet Transfusion | Measured through 24-hours post-operative
  volume in ml/kg
Complete Blood Counts | Pre-specified time points: baseline, ICU admission, 12,24,48,72,96,120 hours post-ultrafiltration.
Total Chest Tube Output | Through study completion, an average of 1 week.
  volume in ml/kg

CONTACTS AND LOCATIONS:
Locations (1):
- IWK Health Centre, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bierer J, Henderson M, Stanzel R, Sett S, Horne D. Subzero balance - simple modified ultrafiltration (SBUF-SMUF) technique for pediatric cardiopulmonary bypass. Perfusion. 2022 Nov;37(8):785-788. doi: 10.1177/02676591211027788. Epub 2021 Jun 18. PMID 34142611
- [Background] Bierer J, Stanzel R, Henderson M, Sett S, Horne D. Ultrafiltration in Pediatric Cardiac Surgery Review. World J Pediatr Congenit Heart Surg. 2019 Nov;10(6):778-788. doi: 10.1177/2150135119870176. PMID 31701831
- [Derived] Bierer J, Stanzel R, Henderson M, Sapp J, Andreou P, Marshall JS, Horne D. Unmasking culprits: novel analysis identifies complement factors as potential therapeutic targets to mitigate inflammation during children's heart surgery. Eur J Med Res. 2024 Dec 19;29(1):601. doi: 10.1186/s40001-024-02156-0. PMID 39696469
- [Derived] Bierer J, Stanzel R, Henderson M, Sett S, Sapp J, Andreou P, Marshall JS, Horne D. Novel inflammatory mediator profile observed during pediatric heart surgery with cardiopulmonary bypass and continuous ultrafiltration. J Transl Med. 2023 Jul 5;21(1):439. doi: 10.1186/s12967-023-04255-8. PMID 37408044